CLINICAL TRIAL: NCT00136539
Title: Neoadjuvant Therapy With Herceptin and Taxol for Stage II/III Breast Cancer
Brief Title: Neoadjuvant Therapy With Herceptin and Taxol for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harold J. Burstein, MD, PhD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Genentech, Inc. (Industry); Bristol-Myers Squibb (Industry); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Harvard Vanguard Medical Associates (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor-Investigator, Harold J. Burstein, MD, PhD, Associate Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-222
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Early Stage Breast Cancer; HER2-positive; HER2-positive breast cancer; Herceptin; Taxol; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: Herceptin — Given intravenously once weekly for 12 weeks prior to surgery.
Drug: Taxol — Given intravenously every 3 weeks (weeks 1, 4, 7, and 10) before surgery.
Drug: Adriamycin — Given every three weeks for 12 weeks after surgery.
Drug: Cytoxan — Given every three weeks for 12 weeks after surgery.

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of administering Herceptin in combination with Taxol (paclitaxel) in the treatment of women with HER2-positive, early stage breast cancer prior to surgery.

DETAILED DESCRIPTION:
Patients will receive Herceptin intravenously once weekly for 12 weeks, and Taxol intravenously every 3 weeks (week 1, week 4, week 7 and week 10).

After 12 weeks of treatment, breast surgery will be performed (either a lumpectomy or a mastectomy).

Once patients have recovered from the surgery, they will receive adriamycin and cytoxan every 3 weeks for 4 cycles (12 weeks total).

After Herceptin and Taxol therapy, tumor assessment will be performed along with an echocardiogram and mammogram.

At the time of surgery, re-assessment of the tumor will be done.

Blood work will be performed on day one of each chemotherapy cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Stage II or III histologically diagnosed breast cancer
* Primary invasive breast cancers that overexpress the HER2/neu oncogene
* Age older than 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of < 1
* White blood cell (WBC) > 4000/mm3
* Platelet count > 100,000/mm3
* Bilirubin < 1 x upper limit of normal (ULN)
* SGOT < 1 x ULN
* Creatinine < 1.5mg/dl
* Normal cardiac function and electrocardiogram (EKG) showing absence of ischemic changes or ventricular hypertrophy

Exclusion Criteria:

* Excisional biopsy, sentinel node dissection or axillary node dissection.
* Prior history of breast cancer unless: diagnosed at least 2 years ago, present cancer is not in a previously irradiated breast, no prior therapy with anthracycline or taxane, no prior high-dose chemotherapy with stem cell or bone marrow transplant.
* Pregnant or breast-feeding women
* Uncontrolled infection
* Active or severe cardiovascular or pulmonary disease
* Peripheral neuropathy of any etiology that exceeds grade 1
* Prior history of malignancy treated without curative intent
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-03; Primary Completion 2006-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the response of HER2-positive breast cancer to treatment with Herceptin and Taxol prior to surgery

SECONDARY OUTCOMES:
To examine the safety of Herceptin and Taxol therapy followed by surgery and chemotherapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts